CLINICAL TRIAL: NCT03607981
Title: Spanish Registry on Spontaneous Coronary Artery Dissection
Acronym: SR-SCAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Spanish Society of Cardiology (Other)
Responsible Party: Principal Investigator, Fernando Alfonso, Head of Cardiology Department, Hospital Universitario de La Princesa, Madrid, Spain, Spanish Society of Cardiology
Other Study IDs: SR-SCAD
Record Dates: First submitted 2018-07-24; First posted 2018-07-31 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Spontaneous Coronary Artery Dissection
MeSH Terms: conditions — Coronary Artery Dissection, Spontaneous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multicenter observational prospective registry, Spanish nationwide-based, of consecutive patients diagnosed with Spontaneous Coronary Artery Dissection (SCAD)

DETAILED DESCRIPTION:
Multicenter prospective registry on patients with diagnosis of Spontaneous Coronary Artery Dissection (SCAD). Spanish nationwide based, the aims of the current registry are:

1. To analyze predisposing factors, potential triggers and associated pathologies of patients presenting with SCAD.
2. To study the clinical and angiographic presentation of these patients.
3. To analyze the value of intracoronary diagnostic techniques (OCT, IVUS) and non-invasive imaging techniques in the diagnosis of this pathology.
4. To better understand the in-hospital clinical evolution and the response to medical treatment or revascularization in these challenging patients, taking into account the angiographic or intravascular imaging morphological characteristics of SCAD and the treatment applied.
5. To analyze its long-term clinical evolution (adverse cardiovascular events, including recurrence of SCAD).
6. To identify those factors directly related to prognostic and risk of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Those consecutive patients with a novel diagnosis of Spontaneous Coronary Artery Dissection (SCAD) that, after careful information, accepted to sign the informed consent form.

Exclusion Criteria:

* Those patients unable to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with a novel diagnosis of Spontaneous Coronary Artery Dissection (SCAD) that meet the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Predictors of adverse events | 3 years
  Clinical, angiographic and imaging predictors of adverse events during follow-up

SECONDARY OUTCOMES:
Predictors of recurrences | 3 years
  Predictors of recurrences of SCAD at follow-up

CONTACTS AND LOCATIONS:
Locations (37):
- Spain (37):
  - Complexo Universitario Hospitalario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Galdakao-Usansolo, Galdakao, Vizcaya
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Complejo Hospitalario Universtario de Albacete, Albacete
  - Hospital General de Alicante, Alicante
  - Hospital Universitario Infanta Cristina, Badajoz
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Puerta del Mar, Cadiz
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital de Cabueñes, Gijón
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Juan Ramón Jiménez, Huelva
  - Complejo Asistencial Universitario de León, León
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario de Torrejon, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital de Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena, Seville
  - Complejo Hospitalario de Toledo, Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alfonso F, Sanz-Ruiz R, Sabate M, Macaya F, Roura G, Jimenez-Kockar M, Nogales JM, Velazquez M, Veiga G, Camacho-Freire S, Moreu J, Pelaez JAF, Perez-Espejo P, Amat-Santos IJ, Diez-Villanueva P, Bastante T, Del Val D, Rivero F, Garcia-Guimaraes M. Clinical Implications of the "Broken Line" Angiographic Pattern in Patients With Spontaneous Coronary Artery Dissection. Am J Cardiol. 2022 Dec 15;185:1-9. doi: 10.1016/j.amjcard.2022.09.017. Epub 2022 Oct 13. PMID 36244863
- [Derived] Garcia-Guimaraes M, Masotti M, Sanz-Ruiz R, Macaya F, Roura G, Nogales JM, Tizon-Marcos H, Velazquez-Martin M, Veiga G, Flores-Rios X, Abdul-Jawad Altisent O, Jimenez-Kockar M, Camacho-Freire S, Moreu J, Ojeda S, Santos-Martinez S, Sanz-Garcia A, Del Val D, Bastante T, Alfonso F; Spanish Registry on SCAD investigators. Clinical outcomes in spontaneous coronary artery dissection. Heart. 2022 Sep 12;108(19):1530-1538. doi: 10.1136/heartjnl-2022-320830. PMID 35410894
- [Derived] Alfonso F, Garcia-Guimaraes M, Alvarado T, Sanz-Ruiz R, Roura G, Amat-Santos IJ, Abdul-Jawad Altisent O, Tizon-Marcos H, Flores-Rios X, Masotti M, Perez-de Prado A, Ferre GF, Ruiz-Poveda FL, Valero E, Portero-Portaz JJ, Diez-Villanueva P, Salamanca J, Bastante T, Rivero F. Clinical implications of arterial hypertension in patients with spontaneous coronary artery dissection. Coron Artery Dis. 2022 Mar 1;33(2):75-80. doi: 10.1097/MCA.0000000000001043. PMID 33878074
- [Derived] Diez-Villanueva P, Garcia-Guimaraes M, Sanz-Ruiz R, Roura G, Macaya F, Barahona Alvarado JC, Tizon-Marcos H, Flores-Rios X, Masotti M, Lezcano-Pertejo C, Cortes C, Fuertes-Ferre G, Becerra-Munoz VM, Lozano Ruiz-Poveda F, Valero E, Portero-Portaz JJ, Vera A, Salamanca J, Alfonso F. Spontaneous coronary artery dissection in old patients: clinical features, angiographic findings, management and outcome. Eur Heart J Acute Cardiovasc Care. 2021 Oct 27;10(8):926-932. doi: 10.1093/ehjacc/zuaa029. PMID 33620451
- [Derived] Diez-Villanueva P, Garcia-Guimaraes MM, Macaya F, Masotti M, Nogales JM, Jimenez-Kockar M, Velazquez M, Lozano I, Moreu J, Avanzas P, Salamanca J, Alfonso F. Spontaneous Coronary Artery Dissection and Menopause. Am J Cardiol. 2021 Jun 1;148:53-59. doi: 10.1016/j.amjcard.2021.02.007. Epub 2021 Feb 20. PMID 33617813
- [Derived] Garcia-Guimaraes M, Bastante T, Macaya F, Roura G, Sanz R, Barahona Alvarado JC, Tizon H, Flores-Rios X, Moreu J, Ojeda S, Nogales JM, Veiga G, Masotti M, Camacho-Freire SJ, Jimenez-Valero S, Jimenez-Kockar M, Lozano I, Gonzalez-Ferreiro R, Velazquez M, Avanzas P, Rivero F, Alfonso F. Spontaneous coronary artery dissection in Spain: clinical and angiographic characteristics, management, and in-hospital events. Rev Esp Cardiol (Engl Ed). 2021 Jan;74(1):15-23. doi: 10.1016/j.rec.2020.04.002. Epub 2020 May 14. English, Spanish. PMID 32418854